CLINICAL TRIAL: NCT00499408
Title: Phase II Trial of Vitamin D and Soy Supplementation for Biochemically Recurrent Prostate Cancer Following Definitive Local Therapy
Brief Title: Vitamin D and Soy Supplements in Treating Patients With Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00000371; P30CA012197 (NIH); CCCWFU-85106; CCCWFU-IRB00000371
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-10

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Vitamin D; Cholecalciferol; Isoflavones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Soy and Vitamin D (Experimental): Patients will receive oral supplementation with both 2,000 IU per day of vitamin D (cholecalciferol) and soy (160 mg per day soy isoflavones). Serum PSA and plasma levels of vitamin D will be assessed monthly. Soy isoflavones levels will be assessed every three months.
  Interventions: Dietary Supplement: Vitamin D; Dietary Supplement: soy

INTERVENTIONS:
Dietary Supplement: Vitamin D — Patients will receive oral supplementation of 2,000 IU per day of vitamin D (cholecalciferol)
  Other Names: cholecalciferol
Dietary Supplement: soy — Patients will receive oral supplementation of soy (160 mg per day soy isoflavones).
  Other Names: isoflavones

SUMMARY:
RATIONALE: Vitamin D and soy extract may be effective in lowering prostate-specific antigen (PSA) levels in patients with recurrent prostate cancer that has not responded to previous treatment.

PURPOSE: This phase II trial is studying how well giving vitamin D together with soy supplements works in treating patients with recurrent prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Test the response of biochemically recurrent prostate cancer to a combination of cholecalciferol (i.e., vitamin D) and soy isoflavones (i.e., soy extract) after failed definitive local therapy as determined by PSA response.

OUTLINE: Patients receive oral cholecalciferol twice daily and a soy supplement (i.e., soy bar or shake) once daily. Treatment continues for 3-12 months in the absence of disease progression or unacceptable toxicity.

Blood samples are obtained at baseline and periodically during study to measure serum PSA, serum calcium, plasma cholecalciferol, and plasma soy isoflavone levels. Blood samples are also analyzed for expression of cholecalciferol receptor, p21, and p27 in peripheral blood lymphocytes as surrogate markers of the actions of cholecalciferol and genistein. Protein expression is assessed by immunoblot analysis of cell lysates as well as quantitative polymerase chain reaction.

Patients complete a toxicity questionnaire once each month to assess for cholecalciferol and soy supplementation toxicities and symptoms of hypercalcemia.

After completion of study therapy, patients are followed every 3 months for 1 year.

ELIGIBILITY:
Inclusion:

* Age > 18 years
* Histologically confirmed adenocarcinoma of the prostate
* Biochemical relapse following definitive therapy by ASTRO criteria (PSA with 3 consecutive rising measurements separated by at least one month) and minimum PSA ≥ 1.0 ng/mL
* PSA doubling time of ≥ 6 months, as demonstrated by 3 PSA measurements obtained ≥ 2 months apart
* No hormonal therapy in 6 months prior to enrollment
* ECOG performance status 0-2
* Life expectancy > 3 months
* At least 2 years since prior definitive radiotherapy
* No concurrent cholecalciferol, calcium, or soy supplements
* Absolute granulocyte count ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Creatinine ≤ 2.0 mg/dL
* Total bilirubin ≤ 2.0 mg/dL
* Calcium > 8.5 mg/dL and < 10.5 mg/dL
* Testosterone ≥ 150 ng/dL

Exclusion:

* No clinically evident brain metastases
* Concurrent cholecalciferol, calcium, or soy supplements
* Concurrent chemotherapy with nonstudy drugs
* Serious medical illness that would limit survival to < 3 months, or psychiatric condition that would preclude giving informed consent
* Other malignancy except nonmelanoma skin cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for the past 5 years
* Active, uncontrolled bacterial, viral, or fungal infection
* Hemorrhagic disorder
* Evidence of metastatic disease by bone scan or CT scan
* History of hypercalcemia
* More History of exposure to other phytotherapeutics, including PC-SPES and Saw Palmetto, within the last year.

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K.C. Balaji, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D and Soy Supplementation: oral supplementation with both 2,000 international units per day of vitamin D (cholecalciferol) and soy (160 milligrams per day soy isoflavones)
Period: Overall Study
Arm/Group | Vitamin D and Soy Supplementation
Started | 26
Completed | 26 (Three patients did not have adequate testing to be evaluable for a response.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vitamin D and Soy Supplementation
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Showing a 50% Reduction in Serum Prostate Specific Antigen(PSA) During Treatment
Time Frame: up to one year
Population: Only 23 participants evaluable for a response.
Measure: Number; unit: participants
Arm/Group | Vitamin D and Soy Supplementation
Number analyzed (Participants) | 23
participants | 0

2. Secondary Outcome: Changes in PSA Slope
Time Frame: up to one year
Population: Data not collected
Arm/Group | Vitamin D and Soy Supplementation
Number analyzed (Participants) | 0

3. Secondary Outcome: Changes in PSA Doubling Time
Time Frame: up to one year
Population: Data not collected
Arm/Group | Vitamin D and Soy Supplementation
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Adverse Events, Grades 1-5
Description: Toxicity will be graded according to the revised NCI Common Terminology Criteria for Adverse Events v 3.0, (CTCAE). Number of events with grade 1-5 will be reported.
Time Frame: up to one year
Measure: Number; unit: events
Arm/Group | Vitamin D and Soy Supplementation
Number analyzed (Participants) | 26
events
  Grade 1 | 93
  Grade 2 | 30
  Grade 3 | 7
  Grade 4 | 0
  Grade 5 | 1

5. Secondary Outcome: Time to Progression
Description: Progression will be defined as a 50% rise in serum PSA compared to the baseline value confirmed on at least two measurements at least two weeks apart.
Time Frame: up to three years
Population: 16 subjects progress out of the 23 evaluable for response.
Measure: Median (Full Range); unit: months
Arm/Group | Vitamin D and Soy Supplementation
Number analyzed (Participants) | 16
months | 10.3 [4 to 35]

ADVERSE EVENTS:
Time Frame: up to 3 years
Arm/Group | Vitamin D and Soy Supplementation
All-Cause Mortality (participants affected / at risk) | 16/26
Serious Adverse Events (participants affected / at risk) | 5/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D and Soy Supplementation (N=26)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
hyperglycemia (Investigations) | 2 (2)
hypoglycemia (Investigations) | 1 (1)
Partial Thromboplastin Time (Investigations) | 1 (1)
Lymphopenia (Investigations) | 1 (1)
Syncope (fainting) (General disorders) | 1 (1)
Skin Infection with high grade neutropenia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D and Soy Supplementation (N=26)
Low WBC (Investigations) | 8 (8)
low Platelets (Investigations) | 6 (6)
Low Hemoglobin (Investigations) | 14 (14)
Nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)
Anorexia (General disorders) | 2 (2)
Alkaline phosphatase (Investigations) | 2 (2)
Creatinine (Investigations) | 3 (3)
"Incontinence, urinary" (General disorders) | 2 (2)
Hypertension (General disorders) | 2 (2)
Taste alteration (General disorders) | 2 (2)
Rigors/chills (General disorders) | 2 (2)
Fatigue (General disorders) | 7 (7)
hyperglycemia (Investigations) | 14 (14)
hypoglycemia (Investigations) | 2 (2)
hypocalcemia (Investigations) | 2 (2)
hyponatremia (Investigations) | 4 (4)
hypoalbuminemia (Investigations) | 2 (2)
hyperbilirubinemia (Investigations) | 2 (2)
hypophosphatemia (Investigations) | 4 (4)
Constipation (Gastrointestinal disorders) | 6 (6)
Pain: Head/headache (General disorders) | 3 (3)
Fever without neutropenia (General disorders) | 2 (2)
Erectile dysfunction (General disorders) | 3 (3)
Urinary frequency/urgency (General disorders) | 14 (14)
Renal/Genitourinary - Other (General disorders) | 2 (2)
Edema: limb (Vascular disorders) | 3 (3)
Dry mouth (General disorders) | 2 (2)
Pain: Abdomen (General disorders) | 4 (4)
Pain: Joint (General disorders) | 2 (2)
Arthritis (non-septic) (General disorders) | 2 (2)
Pain: Back (General disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 4 (4)
Glomerular filtration rate (Investigations) | 2 (2)
"Cholesterol, serum-high" (Investigations) | 2 (2)
Libido (General disorders) | 8 (8)
Lymphopenia (Investigations) | 5 (5)
Pain: Muscle (General disorders) | 6 (6)
Pain: Extremity-limb (General disorders) | 2 (2)
Allergic rhinitis (Skin and subcutaneous tissue disorders) | 11 (11)
"Muscle weakness, generalized or specific area (not due to neuropathy): Extremity-lower" (Musculoskeletal and connective tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
only the most severe of each type of adverse event during treatment was recorded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes